CLINICAL TRIAL: NCT04903743
Title: ULTRASOUND GUIDED POPLITEAL SCIATIC NERVE BLOCK USING BUPIVACAINE ALONE OR COMBINED WITH MAGNESIUM SULFATE FOR DIABETIC FOOT SURGERIES
Brief Title: POPLITEAL SCIATIC NERVE BLOCK FOR DIABETIC FOOT SURGERIES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0106292
Record Dates: First submitted 2021-05-24; First posted 2021-05-26 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Patient
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group B (Placebo Comparator): 28ml of 0.25% bupivacaine and 2ml normal saline
  Interventions: Drug: bupivacaine
- group BM (Active Comparator): received 28 ml of 0.25% bupivacaine and 2 ml magnesium sulfate 10%.
  Interventions: Drug: bupivacaine; Drug: magnesium sulfate

INTERVENTIONS:
Drug: bupivacaine — group B received 28ml of 0.25% bupivacaine and 2ml normal saline
Drug: magnesium sulfate — group BM received 28 ml of 0.25% bupivacaine and 2 ml magnesium sulfate 10%.
  Arms: group BM

SUMMARY:
Popliteal Sciatic nerve block is a regional technique that provides safe and reliable perioperative anesthesia and analgesia of lower leg and foot used in diabetic patients. Different additives have been used with local anaesthetics to achieve dense and prolonged block. Magnesium sulfate possesses analgesic properties owing to its effect on NMDA receptors.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) II or III
* scheduled for diabetic foot surgeries.

Exclusion Criteria:

* Patients who refused the anaesthetic technique,
* whose BMI ≥ 35 kg/ m2,
* unable to properly describe postoperative pain to investigator (dementia, delirium, psychiatric and neurological disorders),
* patients with coagulopathy, skin infection at the site of injection,
* preoperative use of opioid or non-steroidal anti-inflammatory drugs,
* allergy or contraindication to studied medication

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
duration of postoperative analgesia | 24 hours
  evaluate the effects of adding magnesium sulfate to bupivacaine versus bupivacaine alone in popliteal sciatic nerve block with ultrasound guidance for diabetic foot surgeries as regards the duration of postoperative analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- rehab Abd Elaziz, Alexandria, Egypt